CLINICAL TRIAL: NCT02436967
Title: Classification of Carotid Plaque With Computed Tomography With Fast kVp-switching Technique: A Comparison With Histology and 3-Tesla MRI
Brief Title: Classification of Carotid Plaque With Computed Tomography With Fast kVp (Kilovolt Peak)-Switching Technique
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Staffan Holmin, Professor in clinical neuroimaging, Karolinska Institutet
Other Study IDs: SN 020 DECTA
Record Dates: First submitted 2015-03-29; First posted 2015-05-07 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Atherosclerosis; Carotid Stenosis
MeSH Terms: conditions — Atherosclerosis; Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The comparison CT vs histology requires a operated plaque for histology.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Carotid endarterectomy in clinical healthcare. — For the this study itself there is no intervention caused by the extra CT or MRI. The patients are scheduled for surgery as the routine intervention to reduce the risk of a new stroke in clinical practice. The performed extra diagnostic CT and MRI in this study before surgery will compare the vessel wall images with histology regardless of the patients status or medication.

SUMMARY:
Classification of carotid plaque vessel wall changes in carotid stenosis accordingly to AHA classification (American Heart Association)- comparison between histology and CT. The CT is performed with a fast kVp-switching dual energy technique.

To compare the ability to detect iodine contrast enhancement in the carotid plaque compared with 3T MRI with gadolinium.

DETAILED DESCRIPTION:
Patients planned for CEA (carotid endarterectomy) due to carotid stenosis will be examined with one extra CT and MRI before surgery. The CEA specimen is stored in the BiKE-registry (a biobank of operated carotid plaque at the Karolinska Institute). In that registry the patients will be given a personal code which is used to identify the CT, MRI and histology data further on.

Approved by regional ethical review board in Stockholm and local radiation comity at Karolinska University Hospital Solna (Dnr K2435-2014). Informed consent from the participating patients.

ELIGIBILITY:
Inclusion Criteria:

* 50% stenosis (NASCET) or more based on CTA (CT-angiography),
* MRI or US,
* Scheduled for CEA
* 50 years or older,
* Normal kidney function (estimated GFR (glomerular filtration rate) 60 ml/min or more).

Exclusion Criteria:

* Contraindications to iodine contrast media,
* Contraindications to MRI or gadolinium contrast media.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled for CEA (carotid endarterectomy) and volunteer to participate in this study (fulfilling the incl and excl criteria).
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-12; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Classification of the carotid plaque accordingly to AHA classification: Fast kVp-switching dual energy CT with histology | 4 weeks
  The time between radiological examination, surgery and histological analysis is usually approximately 4 weeks

SECONDARY OUTCOMES:
Comparison between the ability to detect contrast enhancement in the carotid plaque: Fast kVp-switching CT vs 3T MRI | 1 week
  The time between fast kVp-switching CT and MRI examinations and reporting is usually approximately 1week.

CONTACTS AND LOCATIONS:
Overall Officials: Staffan Holmin, Professor, Principal Investigator — Dept of Clinical Neuroscience, Karolinska Institutet
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Stary HC, Chandler AB, Dinsmore RE, Fuster V, Glagov S, Insull W Jr, Rosenfeld ME, Schwartz CJ, Wagner WD, Wissler RW. A definition of advanced types of atherosclerotic lesions and a histological classification of atherosclerosis. A report from the Committee on Vascular Lesions of the Council on Arteriosclerosis, American Heart Association. Circulation. 1995 Sep 1;92(5):1355-74. doi: 10.1161/01.cir.92.5.1355. PMID 7648691
- [Result] Cai JM, Hatsukami TS, Ferguson MS, Small R, Polissar NL, Yuan C. Classification of human carotid atherosclerotic lesions with in vivo multicontrast magnetic resonance imaging. Circulation. 2002 Sep 10;106(11):1368-73. doi: 10.1161/01.cir.0000028591.44554.f9. PMID 12221054